CLINICAL TRIAL: NCT02227056
Title: Effect of Methylphenidate on Ecologic Function in Paediatric Acquired Brain Injury Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: loe130007ctil
Record Dates: First submitted 2014-07-01; First posted 2014-08-27 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2018-09

CONDITIONS: Acquired Brain Injury
Keywords: Acquired pediatric brain injury; Methylphenidate; Traumatic brain injury; Cerebrovascular event; Hypoxic ischemic brain injury; Function (ecologic)
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Hypoxia-Ischemia, Brain | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate treatment (Experimental): On three different days each participant will receive Methylphenidate in a dosage of 0.3 milligram/kilo rounded to the nearest full milligram dosage
  Interventions: Drug: Methylphenidate
- Control (No Intervention): On three different days each participant will be re-evaluated without recieveing Methylphenidate.

INTERVENTIONS:
Drug: Methylphenidate — On three different days each participant will receive Methylphenidate in a dosage of 0.3 milligram/kilo rounded to the nearest full milligram dosage
  Other Names: Ritalin
  Arms: Methylphenidate treatment

SUMMARY:
The purpose of this study is to investigate the influence of Methylphenidate in pediatric acquired brain injury population, regarding ecologic (every day) function. It is hypothesized that the function with treatment will improve when compared to function without treatment in the same patient. Improvement is expected by shortening time of execution in each specific task and by reduction of the amount of assistance needed.

DETAILED DESCRIPTION:
Attention deficits in patients with acquired brain injury (ABI) are one of the most common cognitive disorders acquainted. Prevalence of attention deficits after cerebrovascular accident (CVA) varies between 20-58%, and after traumatic brain injury (TBI) may range up to 60% Methylphenidate (MPH) is a central nervous system (CNS) stimulant. In the CNS it increases release and blocks reuptake of dopamine and noradrenalin, resulting in increased synaptic and extracellular concentrations. Methylphenidate (MPH), act at the D1 and α2-adrenergic receptors to facilitate effects on prefrontal cortical modulation of attention and working memory .Methylphenidate has been used effectively and safely for treatment of attention deficit hyperactivity disorder for many decades. The use of Methylphenidate to enhance attention in disorders following TBI has been proposed as "rational pharmacotherapy". It demonstrated improvement in response speed, in adult patients with chronic TBI. In pediatric population suffering Acquired brain injury there are scarce works regarding methylphenidate short or long term efficacy. Since there are scarce reports altogether on Methylphenidate's effect in pediatric Acquired brain injury population and since the studies up to now examined the effectiveness in neuropsychological batteries we find it of interest to examine the effect of Methylphenidate in ecological tasks, thus achieving a better understanding of its possible effect in this subpopulation.

STUDY ASSUMPTIONS:

1. Methylphenidate has a proved safety profile in pediatric population suffering from primary attention deficit hyperactivity disorder or secondary attention deficit hyperactivity disorder .
2. Methylphenidate has positive influence on attentional disorders in pediatric population suffering from Acquired brain injury in subacute and chronic phases.
3. Methylphenidate can enhance function of children with attentional disturbances secondary to Acquired brain injury in different everyday tasks.
4. Methylphenidate can improve learning in pediatric population suffering from secondary attention deficit hyperactivity disorder after Acquired brain injury, during subacute rehabilitation period.

STUDY POPULATION:

The study is designed to include up to 40 children, aged 4-18 years, suffering attentional disturbances secondary to Acquired Brain Injury (CVA, TBI, Anoxic brain injury, Central Nervous System infections). Participants will be children hospitalized (inpatient or outpatient) for rehabilitation in Loewenstein Rehabilitation Center Hospital, with no contraindications for Methylphenidate treatment after their legal guardian gave informed consent for participation.

STUDY METHODS:

1. Before inclusion each participant will undergo:

   1. ECG
   2. A screened computed exam to prove attentional disturbances with the Test of Variables of Attention (TOVA) test.
2. Each participant will be tested on each task twice in two week's period: twice without treatment of Methylphenidate and twice with Methylphenidate treatment.
3. Some participants will be retested after 7-14 days with no further treatment with Methylphenidate, in order to estimate if influence of the drug on function continues with no further treatment.
4. Drug will be given at least an hour and not more than 2.5 hours before being tested.
5. Drug dosage 0.3 milligram/kilo rounded to the nearest full milligram dosage will be given a total of 3 times: once before Test of Variables of Attention (TOVA) exam under Methylphenidate, and two other days while the participant is tested on the different tasks.
6. Testing will be done in two hours of treatment session on different days.
7. Each participant will undergo the following tasks, in a consecutive order:

   1. Dressing -T-shirt. Burden of care graded by scales of The Functional Independence Measure (FIM) or the Functional Independence Measure for Children (WeeFIM) according to age of participant.
   2. Puzzle construction. Two different puzzles to avoid a possibility of learning. Both the same level according to Sheridan's developmental norms.
   3. Mathematical age appropriate working sheet.
   4. Interactive social game such as memory game. On this task each participant will be scored according to number of reminders given for his round or inhibition and his emotional reaction to winning /loosing the game on a scale of 1-5, 1 being appropriate reaction, 5 being highest frustration.
8. The Occupational therapist scoring the child's abilities and amount assistance needed will be blindfolded to the treatment (given or not).

Performance data in each task will be collected with regard to duration for completion, amount of assistance needed, impulsivity, long term and short term attention etc, and statistically analyzed. Each participant (without Methylphenidate treatment) will serve as control to data collected in the same tasks completed under treatment with Methylphenidate .

ELIGIBILITY:
Inclusion Criteria:

1. Male and female.
2. Ages 4-18 years old.
3. No contraindications for Methylphenidate treatment such as hypersensitivity, cardiac disturbances unbalanced seizures etc'.
4. Informed consent given by their legal guardian.
5. Acquired brain injury

Exclusion Criteria:

1. Refusal to participate by either guardian or child.
2. No attentional disturbances in a computed screening exam: "TOVA".
3. Medical contraindications to treatment with Methylphenidate such as short QT syndrome.
4. Side effects due to treatment with Methylphenidate.
5. Under medical treatment of medications enhancing dopamine/ noradrenaline release such as Amantadine.
6. Unable to participate in tasks planned due to severe motor or cognitive disabilities.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2014-01; Primary Completion 2017-01-30 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Measure time (in minutes and seconds) and the amount of assistance needed (number of times each participant needed assistance) to complete the different tasks. | After each task is completed time of the specific task will be recorded. Each participant will be tested 6 times 45 minutes during 3 weeks and will be followed for duration of hospital stay an expected average of 1 month
  Measure the effect of Methylphenidate on function (in everyday tasks like dressing) of children with acquired brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Shaklai, Dr, Principal Investigator — Loewenstein Hospital Rehabilitation Center; Sigal Greenbaum, Master, Study Director — Loewenstein Hospital Rehabiltation Center
Locations (1):
- Loewenstein Rehabilitation Hospital Center, Raanana, Israel

REFERENCES:
- [Background] Willmott C, Ponsford J. Efficacy of methylphenidate in the rehabilitation of attention following traumatic brain injury: a randomised, crossover, double blind, placebo controlled inpatient trial. J Neurol Neurosurg Psychiatry. 2009 May;80(5):552-7. doi: 10.1136/jnnp.2008.159632. Epub 2008 Dec 5. PMID 19060022
- [Background] Hornyak JE, Nelson VS, Hurvitz EA. The use of methylphenidate in paediatric traumatic brain injury. Pediatr Rehabil. 1997 Jan-Mar;1(1):15-7. doi: 10.3109/17518429709060937. PMID 9689233
- [Background] Whyte J, Hart T, Schuster K, Fleming M, Polansky M, Coslett HB. Effects of methylphenidate on attentional function after traumatic brain injury. A randomized, placebo-controlled trial. Am J Phys Med Rehabil. 1997 Nov-Dec;76(6):440-50. doi: 10.1097/00002060-199711000-00002. PMID 9431261
- [Background] Whyte J, Hart T, Vaccaro M, Grieb-Neff P, Risser A, Polansky M, Coslett HB. Effects of methylphenidate on attention deficits after traumatic brain injury: a multidimensional, randomized, controlled trial. Am J Phys Med Rehabil. 2004 Jun;83(6):401-20. doi: 10.1097/01.phm.0000128789.75375.d3. PMID 15166683
- [Background] Wheaton P, Mathias JL, Vink R. Impact of pharmacological treatments on cognitive and behavioral outcome in the postacute stages of adult traumatic brain injury: a meta-analysis. J Clin Psychopharmacol. 2011 Dec;31(6):745-57. doi: 10.1097/JCP.0b013e318235f4ac. PMID 22020351
- [Background] Mahalick DM, Carmel PW, Greenberg JP, Molofsky W, Brown JA, Heary RF, Marks D, Zampella E, Hodosh R, von der Schmidt E 3rd. Psychopharmacologic treatment of acquired attention disorders in children with brain injury. Pediatr Neurosurg. 1998 Sep;29(3):121-6. doi: 10.1159/000028705. PMID 9838263